CLINICAL TRIAL: NCT05167383
Title: A Prospective Randomized Controlled Monocentric Study Evaluating the Impact of Virtual Reality Hypnosis During Labor
Brief Title: Virtual Reality to Reduce Labor Pain
Acronym: VRH4L
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint-Jean, Bruxelles (Other)
Responsible Party: Principal Investigator, Dr. Arnaud Bosteels, Medical doctor, Clinique Saint-Jean, Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRH4L
Record Dates: First submitted 2021-11-06; First posted 2021-12-22 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Labor Pain; Virtual Reality; Hypnosis
Keywords: non-pharmacological analgesia
MeSH Terms: conditions — Labor Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective interventional Randomized Controlled Trial
Who Masked: Investigator
Masking Description: The investigator only gets the anonymized prospective data from the patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention VR group (Active Comparator): . In the VRH group the patients received a 30-minute session of virtual reality hypnosis when in active labor and had access to standard care.
  Interventions: Device: VRH (Virtual Reality Hypnosis); Behavioral: Standard care
- Standard treatment (Placebo Comparator): Patients in the control group received only standard care.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Device: VRH (Virtual Reality Hypnosis) — Hypnosis is delivered as a standardized therapeutic intervention through virtual reality, using a digital sedation software (AQUA ®, Onfomfort SA).
  Arms: Intervention VR group
Behavioral: Standard care — The standard treatment (ST) for labor pain as used in our hospital contains massage, aquatherapy and postural exercises. This is always available for any woman in labor.

SUMMARY:
Background and Goal of Study Labor pain remains an area where different analgesia options are looked for, more specifically non-pharmacological remedies are popular. Hypnosis and virtual reality (VR) have been studied with encouraging results. However, until now, the combination of VR and hypnosis (VRH) has not been assessed during labor, although it has shown promising results in other acute pain areas. The VRH4L study will evaluate the efficacy of Virtual Reality Hypnosis (VRH) in reducing pain during labor. Hypnosis is delivered as a standardized therapeutic intervention through virtual reality, using a digital sedation software (AQUA ®, Oncomfort SA).

For this prospective, interventional parallel group, monocentric randomized controlled trial full term women who were planned for an induction of labor at the St-Jean Hospital in Brussels from March to May 2021 were included. Women with complicated pregnancies and patients with contraindications to VR were excluded.

Patients were randomized in two arms. In the VRH group the patients received a 30-minute session of virtual reality hypnosis when in active labor and had access to standard care. Patients in the control group received only standard care.

Primary outcome was the difference in post intervention pain score between the two arms. Secondary outcomes were the difference in pain score 30 minutes after the intervention, vital signs correlated to pain, satisfaction of the experience, interaction with the midwife and prevalence of side effects. Data was analyzed using the student's T test.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 and ≤ 45 years
2. Pregnant with term gestation
3. Willing to adhere to the rules linked to the use of the VRH headset: turning off mobile phone, visit bathroom in advance, no new visitors and no interference of the partner other than when the woman would ask him so
4. Provision of written informed consent
5. Induced labor

Exclusion Criteria:

1. Complicated pregnancy ( HELLP,…)
2. Scheduled caesarian delivery
3. Receipt of epidural analgesia or opioid painkillers before start active labor phase
4. Low auditory acuity that precludes use of the device
5. Low visual acuity that precludes use of the device
6. Head or face wounds precluding use of the device
7. Schizophrenia
8. Epilepsy
9. Dizziness
10. Non-proficiency in French and/or Dutch (research language)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant woman
Enrollment: 41 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Post interventional pain scores | T1(before intervention) and T3 (directly after intervention)
  Primary outcome was the difference in post intervention pain score between the two arms. Difference in Numerical Rating Scale (0 to 10, where 0 is no pain and 10 is maximum pain) pain scores after the intervention between the VRH and Standard care group.

SECONDARY OUTCOMES:
Pain 30 minutes after intervention | T4 (30 min after intervention)
  Measure of Numerical Rating Scale (0 to 10, where 0 is no pain and 10 is maximum pain) after 30 minutes
Maternal heart rate | T1(before intervention) , T2 (During intervention), T3 (directly after intervention) and T4 (30 min after intervention)
  Measured heart rate during and after intervention as an absolute value.
Nausea | T1(before intervention) , T3 (directly after intervention) and T4 (30 min after intervention)
  Nausea and vomiting scores (0-3, 0 = no nausea, 3= nausea and vomiting))
Satisfaction of the mother | T6 (day 1 postpartum)
  Likert scale (-2,0,2) .-2 is very dissatisfied, 1= dissatisfied, 0= not satisfied, nor dissatisfied, 1= satisfied and 2 is very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Louise Piccart, Dr., Study Chair — Resident Anesthesiologie
Locations (1):
- Clinique Saint-Jean, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Publication of abstract (Poster on the ESA 2021) and Study Report (Paper in the Acta Belgica, end of 2021)
Supporting Information: CSR
Time Frame: end 2021- begin 2022

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT05167383/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT05167383/ICF_001.pdf